CLINICAL TRIAL: NCT04673734
Title: Scan-rescan Reproducibility of Myelin Sensitive MRI Techniques
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-02826; me20Granziera3
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Myelin Integrity
Keywords: Magnetization Transfer Imaging (MTI); Multi-echo Susceptibility-Based imaging (SBI); Myelin Water Imaging (MWI); T1 relaxometry (quantitative T1, qT1); multi-shell diffusion; myelin sensitive MRI techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: myelin sensitive MRI scan — Acquisition of 3 myelin sensitive MRI scans as follows: 1. Two MRI during 1 day; the second after 30 min interval and a repositioning.
  2. One MRI within one week after the first one.
  The total scan time will be ~ 1 hour. T1 maps will be calculated after magnetization-prepared 2 rapid acquisition gradient echoes (MP2RAGE6) acquisition based on a product sequence. Magnetization Transfer (MT) sat maps will be calculated. Quantitative susceptibility mapping (QSM) maps will be reconstructed using an in-house implementation of the structural feature based collaborative reconstruction algorithm (SFCR). For the reconstruction of multi-shell diffusion data, AMICO10 Accelerated Microstructure Imaging via Convex Optimization (AMICO) from diffusion MRI data will be used. Myelin Water Fraction maps will be fitted voxel-wise using a Non-Negative Least Squares fitting.

SUMMARY:
This study is to assess the variation in the measurements of myelin sensitive MRI techniques in both white and grey matter in the brain.

DETAILED DESCRIPTION:
Magnetization Transfer Imaging (MTI) permits the assessment of the integrity of macromolecules in brain tissue, such as myelin and cellular/axonal membrane components.

Multi-echo Susceptibility-Based imaging (SBI) provides quantitative susceptibility maps and T2* maps that - when combined - permit the disentanglement of myelin from iron and various phases of myelin degradation.

Myelin Water Imaging (MWI) quantifies the water trapped between myelin layers by separating the multiple water components in T2 relaxometry data. In fact, the presence of myelin on water pools bound to it provokes a loss in magnetic resonance (MR)-signal coherence, which is more rapid than the one characterizing the water pools located within the axons or in the cytoplasm.

A method based on a spiral acquisition that achieves a myelin-specific signal in clinically compatible scan times is currently applied: T1 relaxometry (quantitative T1, qT1) - which measures the time that a perturbed nuclear spin distribution needs to get back to equilibrium in the longitudinal plane- is sensitive to a number of components of the brain tissue such as myelin, axonal diameter and the overall architectural organization of the brain tissue.

Finally, multi-shell diffusion allows the application of mathematical models of diffusion compartments, which in part are influenced by myelin integrity.

The goal of this study is to assess the stability of these techniques in scan-rescan experiment on 20 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* No neurological or psychiatric disorder

Exclusion Criteria:

* Pregnancy
* Contraindication to MRI (eg, claustrophobia, metallic implants, pacemaker etc).
* Inability to give consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects recruited by public announcements (i.e. advertisement/flyer) on the University Hospital's and the University's notice board
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
analysis of variance between MTI, SBI, MWI, T1 relaxometry and multi-shell diffusion obtained in each subject in each of the 3 scan sessions | 1 hour total scan time (during a time period of max. 1 week)
  statistical analysis of variance between MTI, SBI, MWI, T1 relaxometry and multi-shell diffusion obtained in each subject in each of the 3 scan sessions

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Granziera, Prof. Dr. med., Principal Investigator — Neurologische Klinik und Poliklinik, University Hospital Basel
Locations (1):
- Neurologische Klinik und Poliklinik, University Hospital Basel, Basel, Switzerland